CLINICAL TRIAL: NCT00261911
Title: A 12 Month Study to Assess Safety and Efficacy of Meridia (Sibutramine Hydrochloride Monohydrate) 10 and 15 mg in Obese Adolescents
Brief Title: A Study of Sibutramine in Overweight Adolescents to Assess Weight Loss and Safety.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SB238
Record Dates: First submitted 2005-12-02; First posted 2005-12-06 (Estimated); Last update posted 2007-08-31 (Estimated); Status verified 2007-08

CONDITIONS: Obesity
Keywords: Meridia; Sibutramine; Obesity; Adolescent; BMI
MeSH Terms: conditions — Obesity | interventions — sibutramine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: sibutramine

SUMMARY:
The purpose of this study is to assess the effectiveness of sibutramine on weight loss, reduction in body size and improvement in metabolic risk factors and safety in obese adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Obese adolescent males and females in good general health with a lower limit of inclusion by BMI 2 units above the U.S. weighted mean for the 95th percentile for weight based on age and gender to a BMI of 44 kg/m2, ages 12 to 16 years at randomization. (Efforts should be directed to obtain a study population comprising 50% to 75% females and at least 30% African- Americans across the study. Each site should enroll similar numbers of patients at each age within the 12 to 16 year old age range.)
* Both the patient and legal guardian/parent must be able to communicate meaningfully with the investigator, be legally competent, and provide written informed consent/assent.
* All patients must exhibit sufficient comprehension of written materials to be able to follow diet and exercise recommendations, and to complete written behavioral assessments.
* For females of childbearing potential, a negative pregnancy test will be required prior to study inclusion. Female patients, if sexually active, must be using adequate contraceptive precautions (i.e., oral contraceptives, approved hormonal implant, intrauterine device, diaphragm with spermicide, condom with spermicide). Oral contraceptive use is permitted if used for at least 3 months before starting study medication.
* A serum pregnancy test, which must be negative, is required of all females.
* The patient must have at the screening and baseline visits a mean systolic blood pressure <=130 mm Hg, a diastolic blood pressure <=85 mm Hg, and a pulse rate <=95 beats per minute. Treated hypertensives are allowed in the study if medication has been stable for at least 3 months.

Exclusion Criteria:

* The patient must not have a history of anorexia nervosa.
* The patient must not have a history of clinically significant cardiac disease, congenital heart disease, any clinically significant abnormal cardiac condition, or be known to have a clinically significantly abnormal ECG. Specifically excluded conditions include coronary artery disease, clinically significant cardiac arrhythmias, and congestive heart failure.
* The patient must not have a history of stroke.
* The patient must not have a history of asthma requiring chronic oral corticosteroid therapy. A short course (<7 days) of oral corticosteroid medication is permitted for an acute exacerbation.
* The patient must not have a history of narrow angle glaucoma.
* The patient must not have a history of gallstones unless status post cholecystectomy.
* The patient must not have a history of seizures with the exception of childhood febrile seizure.
* The patient must not have evidence of possible renal dysfunction (creatinine >1.7 mg/dL) or hepatic dysfunction (ALT >50 IU/L, bilirubin >1.0 mg/dL). Patients must not have evidence of active or chronic Hepatitis B or C infection.
* The patient must not be using any of the following medications at any time during the study: monoamine oxidase inhibitors (e.g., furazolidone, phenelzine, procarbazine hydrochloride, selegiline), antidepressant agents (including the use of antidepressant agents for more than 2 weeks during the 90 day period prior to screening), lithium, serotonin reuptake inhibitors, certain opioids (dextromethorphan, meperidine, pentazocine, and fentanyl), prescribed or over-the-counter weight loss agents, centrally acting appetite suppressants, tryptophan, sympathomimetics, serotonergic anti-migraine agents (including sumatriptan succinate, dihydroergotamine, etc.) or any other medication that, in the opinion of the Investigator, may pose harm to the patient, obscure the effects of study medication or interfere with the process of drug absorption, distribution, metabolism, or excretion (i.e., enzyme inducers or enzyme inhibitors).
* Patients may not be taken off an antidepressant for the purposes of entering this study.
* The patient and parent/legal guardian must not have a history of alcohol or drug addiction or substance abuse within the previous two years.
* Patients must not be above the 95th percentile for gender and age for the following categories at Screening, as assessed by the Child Behavior CheckList: "thought problems", "delinquent behavior", "aggressive behavior", or "attention problems".
* The patient must not have a t-score of greater than 65 (significantly above average) for the total Child Depression Inventory score.
* The patient must not have participated in rigorous, structured weight loss programs for more than 2 weeks within the past 6 months prior to screening. Continuing participation in less rigorous programs such as Weight Watchers is allowed; however, the patients must have been a participant for at least 6 months prior to screening to be allowed in the study.
* The patient must not have participated in any investigational drug study within thirty (30) days prior to screening.
* The patient must not have used prescription or OTC (or herbal) weight control medication for more than two (2) weeks during the 180 day period immediately preceding screening. In addition, any such medication is not allowed in the trial.
* The patient must not have previously been a patient/subject in a sibutramine trial or have otherwise used sibutramine.
* Pregnancy
* Pathophysiologic or genetic syndromes associated with obesity (Cushing's syndrome, Turner's syndrome, Prader-Willi syndrome; etc.)
* Diabetes mellitus (FBG greater than or equal to 126 mg/dL)
* Untreated hypothyroidism (TSH greater than 4.0 mU/L for a second generation test)
* Malignancy
* Patient must not have drug screen positive for recreational drugs.
* Coagulopathies or bleeding disorders
* Gastric bypass or other surgical procedure which has the potential to interfere with absorption of study medication, or gastric restrictive surgery.
* Major psychiatric illness in either the patient or patient's legal guardian/parent(s) such as bi-polar disorder, ADD, major depression, bulimia, schizophrenia, psychosis; etc.
* Failure to maintain a minimum level of academic achievement during the previous 6 months prior to screening (patients are excluded if receiving multiple failing grades in school).
* Any other severe medical or psychiatric disorder that precludes participation.

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 498 (Actual)
Dates: Start 2000-07; Study Completion 2002-02

PRIMARY OUTCOMES:
Absolute change in body mass index (BMI) from baseline to endpoint. | 12 months

SECONDARY OUTCOMES:
Percent change from Baseline in BMI | 12 months
Proportions of subjects achieving >= 5% and >=10% BMI and body weight reduction | 12 months
Absolute and percent change from Baseline in waist circumference | 12 months
Body composition (DXA) | 12 months
Lipid and glycemic variables | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Global Medical Information 1-800-633-9110, Study Director — Abbott

REFERENCES:
- [Result] Berkowitz RI, Fujioka K, Daniels SR, Hoppin AG, Owen S, Perry AC, Sothern MS, Renz CL, Pirner MA, Walch JK, Jasinsky O, Hewkin AC, Blakesley VA; Sibutramine Adolescent Study Group. Effects of sibutramine treatment in obese adolescents: a randomized trial. Ann Intern Med. 2006 Jul 18;145(2):81-90. doi: 10.7326/0003-4819-145-2-200607180-00005. PMID 16847290
- [Derived] Daniels SR, Long B, Crow S, Styne D, Sothern M, Vargas-Rodriguez I, Harris L, Walch J, Jasinsky O, Cwik K, Hewkin A, Blakesley V; Sibutramine Adolescent Study Group. Cardiovascular effects of sibutramine in the treatment of obese adolescents: results of a randomized, double-blind, placebo-controlled study. Pediatrics. 2007 Jul;120(1):e147-57. doi: 10.1542/peds.2006-2137. Epub 2007 Jun 18. PMID 17576783